CLINICAL TRIAL: NCT02835079
Title: Treatment Effect of Tamoxifen on Patients With DMD
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Principal Investigator, Talia Dor, MD, Hadassah Medical Organization
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DMDTAM001-HMO-CTIL
Record Dates: First submitted 2016-06-22; First posted 2016-07-15 (Estimated); Last update posted 2022-07-25 (Actual); Status verified 2022-07

CONDITIONS: Duchenne Muscular Dystrophy
Keywords: Duchenne Tamoxifen
MeSH Terms: conditions — Muscular Dystrophy, Duchenne | interventions — Tamoxifen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- open label study (Other): one arm open label study
  Interventions: Drug: Tamoxifen

INTERVENTIONS:
Drug: Tamoxifen

SUMMARY:
Duchenne muscular dystrophy (DMD) is a progressive devastating disease that affects mainly boys, with an incidence of about 1:3,500 live births. The pathology of DMD is a result of non-repaired muscle damage that leads to muscle-tissue replacement by scar tissue, a process known as fibrosis. Currently, there is no effective treatment for the disease. The only therapy offered to these boys are steroids which slightly delayed the disease progression. The boys lose their ability to walk at around the age of 12, and die in the 4th decade of life from severe heart and lung problems.

In this study investigators will test the efficacy of Tamoxifen treatment in ambulatory DMD boys. Tamoxifen is a drug used for palliative treatment of breast cancer patients and has an outstanding safety profile. In addition, Tamoxifen was tested in the past in boys, for other pediatric indications, and showed an excellent safety with no side effects.

Tamoxifen is being tested in this study, as a therapy for DMD, for the following reasons:

(i) it was shown to have anti-fibrotic effect in multiple in-vivo systems; (ii) it assists in the repair of damaged muscles.

In other words, Tamoxifen is expected to have a synergistic effect on DMD patients, due to its dual mechanism of action. Indeed, Tamoxifen was shown to have significant beneficial effects in the mdx mouse model of DMD. Also, a small compassionate cohort of 3 boys, treated for 6 months with Tamoxifen, yielded very encouraging results.

ELIGIBILITY:
Inclusion Criteria:

* Ambulatory

Exclusion Criteria:

* Non Ambulatory

Ages: 5 Years to 16 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 19 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2020-11 (Actual); Study Completion 2020-11 (Actual)

PRIMARY OUTCOMES:
6-minute walk distance (6MWD) | The six minute walk distance will be tested during the 36 months of the trial. For the first 12 months, the 6 minute walk test will be tested every 3 months and for the follow up period of 24 months,will be done every 6 months.
  PT evaluation

SECONDARY OUTCOMES:
North Star assesment(NSAA) | The NSAA will be tested during the 36 months of the trial. For the first 12 months, the NSAA will be tested every 3 months and for the follow up period of 24 months,will be done every 6 months.
  PT evaluation

REFERENCES:
- [Derived] Tsabari R, Simchovitz E, Lavi E, Eliav O, Avrahami R, Ben-Sasson S, Dor T. Safety and clinical outcome of tamoxifen in Duchenne muscular dystrophy. Neuromuscul Disord. 2021 Sep;31(9):803-813. doi: 10.1016/j.nmd.2021.05.005. Epub 2021 Jun 5. PMID 34304968